CLINICAL TRIAL: NCT06678334
Title: Characterization of Transcriptome, Proteome and Metabolome Molecules in Nasal Secretions of Different Subtypes of Chronic Rhinitis
Brief Title: Characteristic Transcriptomic, Proteomic and Metabolomic Molecular Studies of Nasal Secretions From Chronic Rhinitis
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Cheng Lei, Professor, PhD, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2024-SR-580
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collection of plasma and nasal secretions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic rhinitis: In this study, no additional intervention was performed on the patients. Only nasal secretions and blood samples were collected from patients with chronic rhinitis in our hospital.

SUMMARY:
Chronic rhinitis is a common chronic nasal mucosal inflammatory disease. Its clinical symptoms and severity are diverse, mainly including allergic rhinitis, local allergic rhinitis, non-allergic rhinitis with hypereosinophilia syndrome and idiopathic rhinitis. All kinds of rhinitis have clinical symptoms such as nasal congestion, runny nose, sneezing, and nasal itching, but the causes are different. At present, the complicated diagnostic methods of different subtypes of chronic rhinitis are an important factor restricting the improvement of clinical diagnosis and treatment. Based on the found key markers of each subtype of chronic rhinitis, the establishment of a non-invasive classification diagnostic method of chronic rhinitis with nasal secretion as the core is of great practical significance for optimizing the existing clinical diagnosis system and improving the efficiency of clinical diagnosis

DETAILED DESCRIPTION:
To study the characteristic transcriptome, proteome and metabolome molecules of nasal secretions of different subtypes of chronic rhinitis, and to establish a non-invasive diagnostic method for chronic rhinitis based on nasal secretions.Nasal secretions and blood were collected from patients with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. Patients with chronic rhinitis in the Department of Otorhinolaryngology, the First Affiliated Hospital of Nanjing Medical University;
3. Patients who are willing to provide specimens for free to promote the diagnosis of chronic rhinitis.

Exclusion Criteria:

1. Patients received glucocorticoids, immunomodulatory drugs, antihistamines, and other treatments that may affect the study results within the past 1 month.
2. Patients with unstable diseases (including severe asthma) and active immune system diseases;
3. Smoking;
4. Pregnant or lactating women; History of nasal surgery within 5.3 months;

6. Patients with low compliance and refusing to accept specimen and questionnaire collection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients in the First Affiliated Hospital, Nanjing Medical University and volunteering for this study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-06 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
The signature transcriptomic, proteomic, and metabolomic indicators or combinations of nasal secretions of different subtypes of chronic rhinitis | 3 years
  The signature transcriptomic, proteomic, and metabolomic indicators or combinations of nasal secretions of different subtypes of chronic rhinitis, which have high sensitivity and specificity in the diagnosis of a specific chronic rhinitis.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Cheng, PhD, Study Director — The First Affiliated Hospital, Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No
All the individual participant data only available to reasearchers participated in this study